CLINICAL TRIAL: NCT06089083
Title: PROmOting Gynecologic Cancer Patients With Frailty to Achieve Functional Recovery - PROOF Prospective Cohort Study
Brief Title: PROmOting Gynecologic Cancer Patients With Frailty to Achieve Functional Recovery
Acronym: PROOF
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Conquer Cancer Foundation (Other); American Society of Clinical Oncology (Other); National Institute on Aging (NIA) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 23407; NCI-2023-07434 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP)); R03AG088902 (NIH); K12HD001262 (NIH)
Record Dates: First submitted 2023-10-12; First posted 2023-10-18 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Malignant Female Reproductive System Neoplasm; Gynecologic Cancer; Gynecologic Neoplasm
Keywords: Frailty; Risk Factors
MeSH Terms: conditions — Genital Neoplasms, Female; Frailty | interventions — Surveys and Questionnaires; Surgical Procedures, Operative; Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Newly diagnosed gynecologic cancer: Participants will undergo physical function assessments, complete surveys, and medical records every 3 months +/- 4 weeks prior to standard of care surgery (outside of this protocol). After surgery subjects will be followed for at least 3 months +/- 4 weeks for up to one year after diagnosis. Medical record reviews will occur periodically to examine for long-term follow up oncologic outcomes of progression free survival, overall survival, and chemotherapy delays for up to 10 years after enrollment.
  Interventions: Other: Physical function assessment; Other: Self-reported Assessments and Questionnaires; Procedure: Surgery (Standard of Care, Non-Interventional)

INTERVENTIONS:
Other: Physical function assessment — Physical assessments of frailty will be conducted in person.
Other: Self-reported Assessments and Questionnaires — Quality of life questionnaires and self-reported measures will be provided to complete during the course of the study
  Other Names: Questionnaires
Procedure: Surgery (Standard of Care, Non-Interventional) — Surgical data will be reviewed via medical record
  Other Names: Surgical Procedure

SUMMARY:
This study seeks to understand how frailty, a term that describes people who are more vulnerable stressors such as a new medical problem, affects the outcomes and quality of life in adult patients with gynecologic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Assess the risk factors associated with frailty in newly diagnosed gynecologic cancer participants.

SECONDARY OBJECTIVES:

I. Compare primary quality of life endpoint of "healthy days at home" between non-frail and frail participants (primary quality of life endpoint).

II. Compare other perioperative, oncologic, and quality of life outcomes between non-frail and frail participants.

OUTLINE: This is an observational study.

All new patients being evaluated for a new diagnosis of gynecologic cancer by the University of California, San Francisco (UCSF) Gynecologic Oncology service and the Dana-Farber Cancer Institute will be recruited in both the outpatient or inpatient setting. Study participants will be enrolled at the time of diagnosis and followed for up to one year after undergoing surgery for cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or greater
* Undergoing evaluation for a newly diagnosed gynecologic malignancy
* Ability of individual or legal guardian/representative to understand a written informed consent document, and the willingness to sign it

Exclusion Criteria:

* Contraindication to any study-related procedure or assessment
* Does not speak a language for which the consent form and study materials are available

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women undergoing evaluation for a newly diagnosed gynecologic malignancy
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2033-11-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who are categorized as frail | At time of enrollment, 1 day
  The Fried frailty phenotype (FP) assesses physical frailty through five criteria: unintentional weight loss; weakness or poor handgrip strength; self-reported exhaustion; slow walking speed; and low physical activity. Participants who receive a score of >3 will be categorized as 'frail'. Participants who receive a score <=3 will be categorized as Non-frail at time of enrollment.
Demographic risk factors associated with those who screen positive for frailty | At time of enrollment, 1 day
  Demographic risk factors obtained from medical record review (i.e. sex, age, race, ethnicity, cancer type, cancer histology, cancer stage, comorbidities, etc.) will be assessed and analyzed for differences between participants categorized as frail versus non-frail.
Oncologic risk factors associated with those who screen positive for frailty | At time of enrollment, 1 day
  Risk factors determined to be oncologic in nature will be assessed and analyzed for differences between participants categorized as frail versus non-frail.

SECONDARY OUTCOMES:
Mean number of healthy days at home | Up to 10 years
  The number of healthy days at home is defined as healthy days at home is defined as: 365 days minus (1) mortality days, (2) total number of days spent in inpatient, observation, skilled nursing facilities (SNF), rehabilitation, long-term hospital settings, emergency department and will be summarized and used as covariate in analysis.
Mean length of hospital stay | Up to 10 years
  The number of days participants stay in the hospital following standard of care surgery for gynecological cancer will be summarized and used as covariate in analysis.
Percentage of participants readmitted to hospital | Up to 10 years
  Participants with documented re-admission to a hospital following standard of care surgery for gynecological cancer will be summarized and used as a covariate in analysis.
Percentage of participants with reported surgical complications | Up to 10 years
  Participants with documented peri-operative complications following standard of care surgery for gynecological cancer will be summarized and used as a covariate in analysis.
Mean time to initiation of standard of care chemotherapy | Up to 10 years
  The median number of days following standard of care surgery for gynecological cancer to first standard of care chemotherapy initiation will be summarized and used as a covariate in analysis.
Median Progression Free Survival (PFS) | Up to 10 years
  Progression free survival is defined as the time from date of diagnosis to date of radiographic progression, and/or doubling of cancer antigen 125 (CA-125) from baseline.
Median Overall Survival (OS) | Up to 10 years
  Overall survival as defined by days from date of diagnosis to date of death, or study completion whichever occurs first.
Mean number of treatment delays | Up to 10 years
  Chemotherapy delays is defined by the number of chemotherapy infusions that are delayed due for medical purposes and the total number of days infusions are delayed for will be summarized and used as a covariate in analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Cham, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No